CLINICAL TRIAL: NCT04794296
Title: Recommendations for the Treatment of Children With Acute Lymphoblastic Leukemia in the GFAOP
Acronym: LALGFA2019
Status: Recruiting | Type: Observational
Sponsor: French Africa Pediatric Oncology Group (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: LAL-GFAOP2019
Record Dates: First submitted 2021-01-22; First posted 2021-03-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Childhood ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The LALGFA2019 Recommendations redefine the standard risk criteria and propose to introduce anthracycline induction in so-called high-risk forms (LAL line T and LAL line B with leukocytosis greater than or equal to 50 G/L or in children less than 1 year of age or more than 10 years of age) as well as Endoxan and Methotrexate in high dose consolidation.

DETAILED DESCRIPTION:
A few studies conducted in developing countries confirm that it is possible to significantly improve the prognosis of children with Acute Lymphoblastic Leukemia (ALL) provided that the centres can benefit from a precise and adapted protocol and logistical support.

The GFAOP has been working with units for the past 20 years and this is the second study put in place by the group for the treatment of LAL. The initial study was a feasibility study with the treatment of standard risk LAL. This study GFALAL2019 aims to include both standard and high-risk forms of LAL.

With this study it is hoped to:

1. Ensure the feasibility of these recommendations.
2. To show that the correct application of the therapeutic recommendations will result in a complete remission rate (CR) close to 85% at the end of the induction treatment.
3. The survival without relapse of patients in RC will be close to 65% at 5 years.

ELIGIBILITY:
Inclusion Criteria:

Children 0 to 18 ALL first diagnosis No prior chemotherapy Cytology FAB L1 or L2

-

Exclusion Criteria:

ALL L3 (Burkitt) ALL previously treated with chemotherapy Trisomy 21

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 0 to 18 years of age presenting for treatment in any of the unit selected to carry out the recommandations
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of these recommendations | This can be initially reviewed after the first 2 years and will be evaluated at the end for the community.
  Availability of drugs. This is part of the project as we are working with Low or low to Middle Income countries.
Correct application of therapeutic recommendations | 5 weeks
  Availability of drugs and adherence to protocol: Some centers may at times have to find locally the chemiotherapy for application of the protocol. The capacity of the units to do this is alos being studied. By looking at why treatment was not given. Was it because of lack of discipline regarding the attendance at the units for treatment, transport, accommodation, or medication not available ?
Complete Remission Rate (CR) close to 85% after induction | J 34 or j42 post start of induction treatment for all children studied.
  Evaluation of the CR j34 or J42 depending on the risk level High or standard.
Ability to follow treatment: | 5 weeks
  The number of children who stop treatment without the consent of the doctor.
Outcome | 5 years
  The vital status at the end of the first line of treatment.

SECONDARY OUTCOMES:
Survival without relapse of patients | first evaluation starts in 2026 so that enough time has elapsed to evaluate.
  the number of children in complete remission without relapse at the end of treatment .

CONTACTS AND LOCATIONS:
Locations (3):
- CHU de Treichville à ABIDJAN, Abidjan, Côte d’Ivoire
- CHU Donka 030 BP 554, Conakry, Guinea
- Hôpital Aristide Le Dantec, Avenue Pasteur,, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided